CLINICAL TRIAL: NCT00809588
Title: A Phase IB Study of Vaccination With Autologous, Lethally Irradiated Melanoma Cells Engineered by Adenoviral Mediated Gene Transfer to Secrete Human Granulocyte-Macrophage Stimulating Factor
Brief Title: Vaccination With Autologous, Lethally Irradiated Melanoma Cells Engineered by Adenoviral Mediated Gene Transfer to Secrete Granulocyte-Macrophage Stimulating Factor (GMSF)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, F. Stephen Hodi, MD, Melanoma Disease Center Director, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-218
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Melanoma
Keywords: vaccination; GM-CSF; autologous; irradiated
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Melanoma Vaccine (Experimental): GM-CSF Vaccine
  Interventions: Biological: Autologous, lethally irradiated melanoma cells

INTERVENTIONS:
Biological: Autologous, lethally irradiated melanoma cells — Engineered to secrete human granulocyte-macrophage stimulating factor. Given on days 1, 8, 15, 29 and every two weeks after until the supply of vaccine has run out

SUMMARY:
The purpose of this study is to see if the proposed therapy will delay or stop the progression of the participants skin cancer. This study is being done because there are currently no treatments which have been shown convincing to treat disease which has progressed. This research study is designed to evaluate the immunologic effects and clinical side effects of giving vaccines to patients that are made from their own skin cancer cells.

DETAILED DESCRIPTION:
* The vaccines created from the participants melanoma cells are scheduled to be given to the participants on days 1, 8, 15, 29 and every two weeks after until the supply of vaccine has run out. The amount of vaccine is dependent on the total amount of cells yielded when the tumor is processed and treated. It is hoped that participants will receive at least six vaccines.
* The vaccines will be administered in two injections that will be placed underneath the participants skin. The two injections will be given at the same place on the body.
* If tumor sample yields enough cells, participants will also receive an injection of non-transduced irradiated melanoma cells. The purpose of this is to measure the amount of reaction of the participants immune system occuring created by the vaccine.
* If either the vaccine site or DTH placement site has shown a reaction, a punch-biopsy will be taken. This will consist of a small piece of skin tissue removed under local anesthesia.
* With vaccine #5, participants will receive a second DTH injection. Two days after the vaccine and DTH injection, punch biopsies will be taken of both sites.
* At week 10 of treatment (or earlier if necessary), participants will undergo a chest, abdomen and pelvic CT scan. The physician may also have participants undergo a brain MRI if indicated at this time.

ELIGIBILITY:
Inclusion Criteria:

* Stage III patients must have: A) Histologically documented melanoma B) Lymphadenopathy of at least 2cm in greatest diameter by physical exam or CT scan in a region draining a known or suspected primary melanoma or in transit metastatic disease of at least 2cm in greatest diameter by physical exam or CT in a region draining a known primary melanoma C) refused, not eligible, or failed adjuvant therapy with high dose a-interferon D) must be able to have all measurable disease removed at time of tumor harvest
* Stage IV patients must have histologically documented metastatic melanoma
* ECOG Performance Status 0 or 1
* Estimated life expectancy of 6 months or greater
* 18 years of age or older
* Signed Informed Consent
* Greater than 4 weeks from any chemotherapy, radiotherapy, immunotherapy, or systemic glucocorticoid therapy
* Greater than 6 months since bone marrow or peripheral blood stem cell transplant

Exclusion Criteria:

* Uncontrolled active infection
* Pregnancy or nursing mothers
* Evidence of infection with Human Immunodeficiency Virus, Hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2003-10-16 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
To determine the doses of lethally irradiated, autologous melanoma cells engineered by adenoviral mediated gene transfer to secrete CM-CSF that can be manufactured in stage III melanoma patients. | 7 years

SECONDARY OUTCOMES:
To determine the safety and biologic activity of vaccination with lethally irradiated, autologous melanoma cells engineered by adenoviral mediated gene transfer to secrete GM-CSF | 7 years
To determine the two-year survival of stage IV melanoma patients vaccinated with lethally irradiated, autologous melanoma cells engineered by adenoviral mediated gene transfer to secrete GM-CSF | 7 years
To determine more fully the safety and biologic activity of vaccination with lethally irradiated, autologous melanoma cells engineered by adenoviral mediated gene transfer to secrete GM-CSF in stage IV melanoma patients | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: F. Stephen Hodi, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts